CLINICAL TRIAL: NCT04536090
Title: An Open-Label Randomized Study of Isoquercetin (IQC-950AN) Plus Standard of Care Versus Standard of Care Only for the Treatment of 2019 Novel Coronavirus Disease (COVID-19)
Brief Title: Study of Isoquercetin (IQC-950AN) Plus Standard of Care Versus Standard of Care Only for the Treatment of COVID-19
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Never started
Sponsor: Institut de Recherches Cliniques de Montreal (Other)
Collaborators: Pharmascience Inc. (Industry); SCiAN Services, Inc. (Unknown); Quercis Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRCM-IQC-001
Record Dates: First submitted 2020-08-31; First posted 2020-09-02 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: COVID-19
Keywords: Isoquercetin; Quercetin; Antiviral Agents
MeSH Terms: conditions — COVID-19 | interventions — isoquercitrin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Isoquercetin (IQC-950AN) (Experimental): 1000 mg Isoquercetin b.i.d. on day 1, then 500 mg Isoquercetin b.i.d. for 27 more days, plus standard of care (as defined below)
  Interventions: Drug: Isoquercetin (IQC-950AN)
- Standard of care (No Intervention): This arm will receive standard of care based on national guidelines. This may change as new information regarding best practice emerges.

INTERVENTIONS:
Drug: Isoquercetin (IQC-950AN) — Isoquercetin will be administered by mouth twice daily for 28 days
  Other Names: IQC-950AN
  Arms: Isoquercetin (IQC-950AN)

SUMMARY:
This is an open-label, randomized, multi-centre study where hospitalized subjects will be randomized in a 2:1 ratio to receive Isoquercetin (IQC-950AN) in addition to standard of care or standard of care only for 28 days following confirmation of a COVID-19 infection.

DETAILED DESCRIPTION:
The primary purpose of this randomized study will be to evaluate the effect of Isoquercetin (IQC-950AN) treatment on disease progression (defined as ≥ 6 on the World Health Organization (WHO) clinical progression scale) when given to subjects with confirmed COVID-19 in addition to standard of care. The secondary purpose of this study is to evaluate the effect of Isoquercetin (IQC-950AN) treatment on the reduction of severe acute respiratory coronavirus 2 (SARS-CoV-2) viral titers in these subjects and their recovery. In addition, certain parameters which may help elucidate the mechanism of action (sLDLR, PCSK9, sACE2, D-dimers and CRP) will be followed. The safety of Isoquercetin (IQC-950AN) will be evaluated at each visit. Subjects will be randomized to receive treatment for 28 days and then will return 30 days following the discontinuation of treatment for a final safety visit.

The results of this study will be used to design an adequately powered randomized controlled pivotal study to evaluate the efficacy and safety of Isoquercetin (IQC-950AN) in all or a subset of subjects with confirmed COVID-19.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must exhibit symptoms of COVID-19 disease at screening;
2. Patients must be 18 years of age or older, of either gender;
3. Patients must have a documented SARS-CoV-2 RNA-positive test virus within 3 days prior to randomization;
4. Patients must be admitted (or under observation to be admitted) to a controlled facility or hospital to receive standard-of-care for COVID-19 disease;
5. Patient's health status must be 3 (if hospitalized for comorbidities), 4, or 5 on the WHO clinical progression scale defined as hospitalized moderate disease (no oxygen therapy or oxygen by mask or nasal prongs);
6. If female, must be either post-menopausal (one year or greater without menses), surgically sterile, or, for female subjects of child-bearing potential who are capable of conception, must be: practicing a highly effective method of birth control during the study and through 30 days after the last dose of the study medication.
7. Patients must have the ability to understand and give informed consent, which can be verbal with a witness, according to local requirements;
8. Patients deemed capable of adequate compliance including attending scheduled visits for the duration of the study;
9. Patients must be able to swallow the study drug capsules

Exclusion Criteria:

1. Patients with a history of allergy or anaphylaxis to ingredients in Isoquercetin (IQC-950AN) including known intolerance of niacin or ascorbic acid or known glucose-6-phosphate dehydrogenase (G6PD) deficiency;
2. Patients with known chronic kidney disease with estimated creatinine clearance < 50 mL/minute or need for dialysis;
3. Patients receiving an intensified dose regimen of low molecular weight heparin (LMWH) or unfractionated heparin (defined as doses of LMWH or unfractionated heparin greater than those approved for thromboprophylaxis) or dual antiplatelet therapy;
4. Patients who are severely hypotensive defined as needing hemodynamic pressors to maintain blood pressure;
5. Patients with moderate or severe thrombocytopenia (platelet count <100 × 10⁹/L);
6. Patients who are breast-feeding an infant or child;
7. Patients who are pregnant or unwilling to use an appropriate form of contraception, except for heterosexual celibacy
8. Any other condition that, in the opinion of the investigator, may adversely affect the patient's ability to complete this study or its measures, or pose a significant risk to the patient;
9. Any reason the investigator suspects that data collected from this patient would be incomplete or of poor quality

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Disease Progression | 28 days
  Disease progression is defined as WHO Clinical Progression Scale ≥6, at any time between Day 1 and Day 28

SECONDARY OUTCOMES:
Changes in viral load from baseline to end of treatment - Mean viral load | 28 days
  Viral load of SARS-CoV-2 RNA (# of viral copies) assessed by quantitative reverse transcription polymerase chain reaction (qRT-PCR)
Changes in viral load from baseline to end of treatment - Area under the viral load vs. time profiles | 28 days
  Viral load of SARS-CoV-2 RNA (# of viral copies) assessed by quantitative reverse transcription polymerase chain reaction (qRT-PCR)
Changes in viral load from baseline to end of treatment - Time profile of viral load | 28 days
  Viral load of SARS-CoV-2 RNA (# of viral copies) assessed by quantitative reverse transcription polymerase chain reaction (qRT-PCR)
Changes in viral load from baseline to end of treatment - Percentage of patients that are viral negative | 28 days
  Defined as below the level of quantitation of the assay (qRT-PCR). Viral load of SARS-CoV-2 RNA (# of viral copies) assessed by quantitative reverse transcription polymerase chain reaction (qRT-PCR)
Disease Recovery | 28 days
  Disease recovery is defined as WHO Clinical Progression Scale score of ≤2
Change in WHO Clinical Progression Scale score | 28 days
  Change in score from baseline to day 28
Incidence of all-cause mortality | 30 days
  All-cause mortality calculated at Day 30
Progression to supplementary oxygen requirement | 14 days
  If the patient required supplementary oxygen during hospitalization
Incidence of mechanical ventilation | 14 days
  If the patient required mechanical ventilation during hospitalization
Incidence of ICU admission | 14 days
  If the patient was admitted to ICU
Time to hospital discharge | 29 days
  Length of time in hospital prior to being discharged
Changes in serum C reactive protein levels (CRP) | 29 days
  Changes in serum CRP levels
Changes in D-dimer levels | 29 days
  Changes in D-dimer levels
Changes in soluble low-density lipoprotein receptor (sLDLR) expression and proprotein convertase subtilisin/kexin type 9 (PCSK9) and soluble angiotensin converting enzyme 2 (sACE2) levels | 29 days
  Changes in sLDLR expression, and PCSK9 and sACE2 levels
Changes in LDL-cholesterol | 29 days
  Changes in LDL-cholesterol
Changes in creatinine | 29 days
  Changes in creatinine
Changes in liver enzymes | 29 days
  Changes in liver enzymes

CONTACTS AND LOCATIONS:
Overall Officials: Michel Chrétien, FRS MD FRCP©, Study Director — Montreal Clinical Research Institute

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] WHO Working Group on the Clinical Characterisation and Management of COVID-19 infection. A minimal common outcome measure set for COVID-19 clinical research. Lancet Infect Dis. 2020 Aug;20(8):e192-e197. doi: 10.1016/S1473-3099(20)30483-7. Epub 2020 Jun 12. PMID 32539990